CLINICAL TRIAL: NCT03156829
Title: Effectiveness of Cortisone Injection and Splinting for Trigger Finger: A Prospective Randomized Controlled Trial
Brief Title: Effectiveness of Cortisone Injection and Splinting for Trigger Finger
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 10016406
Record Dates: First submitted 2017-05-08; First posted 2017-05-17 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Trigger Finger
Keywords: splinting; steroid; cortisone; trigger digit
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Splints; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Splint alone (Experimental)
  Interventions: Other: Splint
- Cortico-steroid alone (Experimental)
  Interventions: Drug: Betamethasone
- Splint and cortico-steroid combined (Experimental)
  Interventions: Combination Product: Splint + Cortico-steroid injection

INTERVENTIONS:
Other: Splint — Custom made splint
  Arms: Splint alone
Drug: Betamethasone — Corticosteroid Injection Brand name of the drug: Celestone Soluspan Dosage: 6 mg/ml
  Arms: Cortico-steroid alone
Combination Product: Splint + Cortico-steroid injection — Splint + Cortico-steroid injection given in combination
  Arms: Splint and cortico-steroid combined

SUMMARY:
Trigger finger has a prevalence rate of up to 3%. There are many approaches available to manage this condition. While corticosteroid injection is widely accepted as the most common first-line treatment, its superiority over splint treatment has not been established. This study aims to test the effectiveness of cortisone injections, splint and cortisone+splint to resolve symptoms.

DETAILED DESCRIPTION:
BACKGROUND:

Multiple approaches, such as nonsteroidal anti-inflammatory medication (NSAIDs), splinting, percutaneous surgery, and open surgery, are available for managing trigger finger, blind corticosteroid injection has been widely accepted as the most common first-line treatment (Castellanos 2015). Splinting is helpful in reducing symptoms, is relatively inexpensive and has a low risk of complications, however, no concrete evidence exists to support the role of splinting in patients presenting with trigger finger (Tarbhai 2012). Surgical intervention is the most effective treatment; however, it is associated with higher risks and loss of time from work (Nimigan 2006). Corticosteroid injection is considered the most effective treatment to resolve symptoms in nondiabetic patients, as the success rate is slightly lower in patients with diabetes (Nimigan 2006). Although there are few studies suggesting effectiveness of cortisone injections and splinting for patients with trigger finger. There is lack of consensus on whether cortisone injections and splinting are effective on their own or in combination to resolve patient symptoms in the long term.

OBJECTIVE:

The objective is to prospectively compare the effectiveness of cortisone injections, splint and cortisone+splint for complete resolution of symptoms for the entirety of the follow-up period.

STUDY DESIGN AND METHODOLOGY:

This is a randomized controlled trial. On receipt of consent, the subjects will be screened for eligibility criteria and informed about the study by their surgeon or their delegate, Katrina Munro who is a research assistant working on this project. They will be informed that if they choose to participate, they will be randomized to receive either a splint, corticosteroid injection or both. Side effects will be explained. In keeping with standard ethical procedures, patients will be informed about confidentiality, that their care will not be affected by their choice, and their rights to withdraw consent at any time. Upon receiving verbal consent, patients will sign the consent form approved by the institutional/ ethics review board. Once a patient has consented, block randomization will occur according to the following stratification variables: A.Severity Grade 1 (pain/history of catching) and Grade 2 (demonstrable catching, can actively extend) Grade 3 (demonstrable locking, requiring passive extension) B. Diabetes (y/n)

DATA ANALYSIS:

Statistical Package for Social Sciences for Windows software (SPSS version 23, IBM SPSS Inc., Chicago, Ill., USA) for Windows (Microsoft) will be used for statistical analyses. Variables will be expressed as mean and range or mean ± SD, as appropriate. Univariate analysis will be used to compare clinical, and demographic data between study groups, including independent t-test for continuous variables and chi square test for categorical variables. General linear models with repeated measures of ANOVA and mixed model ANOVA will be used to examine the change in outcomes within and between the participant groups respectively. Non-parametric tests will be employed when applicable. Logistic and linear multivariate regression analysis will be used to examine binary and continuous outcome variables respectively, controlling for confounding variables.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature adults
2. Symptom duration of at least 3 months
3. Diagnosis of trigger finger: based on history of triggering and physical examination (pain over the flexor tendon, tenderness or nodule over the A1 pulley, stiffness, and reproducible locking or triggering).
4. Green's Grade 1-3 (Green's Classification to Grade the Severity of Trigger Finger)

Exclusion Criteria:

1. Congenital trigger thumb
2. Green's Grade 4 (fixed flexion contracture)
3. Previous treatment for trigger finger (injection or surgery)
4. Allergy to cortisone
5. Multiple digits (>2 digits)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Resolution of symptoms | 6 week
  complete relief/partial relief/no relief
Resolution of symptoms | 3 month
  complete relief/partial relief/no relief
Resolution of symptoms | 6 month
  complete relief/partial relief/no relief
Resolution of symptoms | 1 year
  complete relief/partial relief/no relief

SECONDARY OUTCOMES:
Patients' experiences with the splint - Compliance | 6 week
  1 poor 2 fair 3 good 4 very good 5 excellent
Patients' experiences with the splint - Compliance | 3 month
  1 poor 2 fair 3 good 4 very good 5 excellent
Patients' experiences with the splint - Compliance | 6 month
  1 poor 2 fair 3 good 4 very good 5 excellent
Patients' experiences with the splint - Compliance | 1 year
  1 poor 2 fair 3 good 4 very good 5 excellent
Patients' experiences with the splint - Comfort | 6 week
  1 very uncomfortable 2 uncomfortable 3 neither 4 comfortable 5 comfortable
Patients' experiences with the splint - Comfort | 3 month
  1 very uncomfortable 2 uncomfortable 3 neither 4 comfortable 5 comfortable
Patients' experiences with the splint - Comfort | 6 month
  1 very uncomfortable 2 uncomfortable 3 neither 4 comfortable 5 comfortable
Patients' experiences with the splint - Comfort | 1 year
  1 very uncomfortable 2 uncomfortable 3 neither 4 comfortable 5 comfortable
Patients' experiences with the splint - Ease of use | 6 week
  1 Very difficult 2 Difficult 3 Neutral 4 Easy to use 5 Very easy to use
Patients' experiences with the splint - Ease of use | 3 month
  1 Very difficult 2 Difficult 3 Neutral 4 Easy to use 5 Very easy to use
Patients' experiences with the splint - Ease of use | 6 month
  1 Very difficult 2 Difficult 3 Neutral 4 Easy to use 5 Very easy to use
Patients' experiences with the splint - Ease of use | 1 year
  1 Very difficult 2 Difficult 3 Neutral 4 Easy to use 5 Very easy to use
Pain (Visual analogue scale) | 6 week
  on a scale ranging from "No pain" to "Pain as bad as it could possibly be")
Pain (Visual analogue scale) | 3 month
  on a scale ranging from "No pain" to "Pain as bad as it could possibly be")
Pain (Visual analogue scale) | 6 month
  on a scale ranging from "No pain" to "Pain as bad as it could possibly be")
Pain (Visual analogue scale) | 1 year
  on a scale ranging from "No pain" to "Pain as bad as it could possibly be")
Incidence of Triggering: Number of times finger 'catches' with 10 repeated grip attempts | 6 weeks
  Number of times
Incidence of Triggering: Number of times finger 'catches' with 10 repeated grip attempts | 3 month
  Number of times
Incidence of Triggering: Number of times finger 'catches' with 10 repeated grip attempts | 6 month
  Number of times
Incidence of Triggering: Number of times finger 'catches' with 10 repeated grip attempts | 1 year
  Number of times
Incidence of Triggering: Severity (on Greens Grading Criteria) | 6 week
  Grade 1: Pain/history of catching Grade 2: Demonstrate catching, but can actively extend the digit Grade 3: Demonstrate locking, requiring passive extension Grade 4: Fixed flexion contracture
Incidence of Triggering: Severity (on Greens Grading Criteria) | 3 month
  Grade 1: Pain/history of catching Grade 2: Demonstrate catching, but can actively extend the digit Grade 3: Demonstrate locking, requiring passive extension Grade 4: Fixed flexion contracture
Incidence of Triggering: Severity (on Greens Grading Criteria) | 6 month
  Grade 1: Pain/history of catching Grade 2: Demonstrate catching, but can actively extend the digit Grade 3: Demonstrate locking, requiring passive extension Grade 4: Fixed flexion contracture
Incidence of Triggering: Severity (on Greens Grading Criteria) | 1 year
  Grade 1: Pain/history of catching Grade 2: Demonstrate catching, but can actively extend the digit Grade 3: Demonstrate locking, requiring passive extension Grade 4: Fixed flexion contracture
Patient Rated Wrist Hand Evaluation (PRWHE) - self reported questionnaire | 6 week
  on a scale of 0 (good) to 100 (poor)
Patient Rated Wrist Hand Evaluation (PRWHE) - self reported questionnaire | 3 month
  on a scale of 0 (good) to 100 (poor)
Patient Rated Wrist Hand Evaluation (PRWHE) - self reported questionnaire | 6 month
  on a scale of 0 (good) to 100 (poor)
Patient Rated Wrist Hand Evaluation (PRWHE) - self reported questionnaire | 1 year
  on a scale of 0 (good) to 100 (poor)
Grip Strength (Affected hand) | 6 week
  Kilogram (Kg)
Grip Strength (Affected hand) | 3 month
  Kilogram (Kg)
Grip Strength (Affected hand) | 6 month
  Kilogram (Kg)
Grip Strength (Affected hand) | 1 year
  Kilogram (Kg)
Grip Strength (Un-affected hand) | 6 weeks
  Kilogram (Kg)
Grip Strength (Un-affected hand) | 3 month
  Kilogram (Kg)
Grip Strength (Un-affected hand) | 6 month
  Kilogram (Kg)
Grip Strength (Un-affected hand) | 1 year
  Kilogram (Kg)
Range of motion (Extensor lag) | 6 weeks
  degrees
Range of motion (Extensor lag) | 3 month
  degrees
Range of motion (Extensor lag) | 6 month
  degrees
Range of motion (Extensor lag) | 1 year
  degrees

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Grewal, MD, Principal Investigator — Schulich School of Medicine and Dentistry\Surgery
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castellanos J, Munoz-Mahamud E, Dominguez E, Del Amo P, Izquierdo O, Fillat P. Long-term effectiveness of corticosteroid injections for trigger finger and thumb. J Hand Surg Am. 2015 Jan;40(1):121-6. doi: 10.1016/j.jhsa.2014.09.006. Epub 2014 Oct 14. PMID 25443167
- [Background] Tarbhai K, Hannah S, von Schroeder HP. Trigger finger treatment: a comparison of 2 splint designs. J Hand Surg Am. 2012 Feb;37(2):243-9, 249.e1. doi: 10.1016/j.jhsa.2011.10.038. Epub 2011 Dec 20. PMID 22189188
- [Background] Nimigan AS, Ross DC, Gan BS. Steroid injections in the management of trigger fingers. Am J Phys Med Rehabil. 2006 Jan;85(1):36-43. doi: 10.1097/01.phm.0000184236.81774.b5. PMID 16357547